CLINICAL TRIAL: NCT02174575
Title: Effects of Different Inhalational Anesthetic Agents on the Incidence of Clinical and Subclinical Acute Kidney Injury After Liver Resection Surgery: a Pilot Study
Brief Title: Anesthetic Agents and Acute Kidney Injury After Liver Resection Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: I retired my post before enrollment
Sponsor: Tokyo Medical and Dental University (Other)
Responsible Party: Principal Investigator, Koshi Makita, MD, Professor, Tokyo Medical and Dental University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TMDU-1490
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma; Hepatoma; Cholangiocarcinoma; Gallbladder Neoplasms
Keywords: Hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Active Comparator): Patients are randomized into 2 groups (Desflurane group and Sevoflurane group) depending on the anesthetic agents administered during anesthesia.
  Interventions: Drug: Sevoflurane
- Desflurane (Active Comparator): Patients are randomized into 2 groups (Desflurane group and Sevoflurane group) depending on the anesthetic agents administered during anesthesia.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane is administered during anesthesia in Sevoflurane group.
  Arms: Sevoflurane
Drug: Desflurane — Desflurane is administered during anesthesia in Desflurane group.
  Arms: Desflurane

SUMMARY:
* It has been shown that patients who undergo liver resection surgery are at high risk for postoperative acute kidney injury (AKI).
* Sevoflurane may increase the risk for postoperative AKI because of production of compound-A.
* Therefore, we have planned to investigate the effects of different anesthetic agents on postoperative renal function.
* Patients undergoing liver resection surgery are randomized into 2 groups.
* One of the groups receives sevoflurane and the other group receives desflurane.
* Blood and urine specimen are sampled both pre- and postoperatively, and several biomarkers are compared between the groups.

DETAILED DESCRIPTION:
1. Design

   - This is a randomized, observer-blinded, controlled trial.
2. Study objectives and hypothesis

   - The aim of this study is to prove the hypothesis that desflurane is safer than sevoflurane in terms of the association with postoperative acute kidney injury (AKI) after liver resection surgery.
3. Inclusion and exclusion criteria

   * Inclusion criteria: Forty adult patients (20 patients in each group) who are planned to undergo liver resection surgery are included.
   * Exclusion criteria: Patients who undergo less invasive liver resection surgery under thoracoscopy or laparoscopy are excluded. Patients with chronic kidney disease, or allergic to any anesthetic agents used in the study (e.g., desflurane, sevoflurane, propofol, remifentanil, rocuronium) are also excluded.
4. Outcome definition

   - AKI is diagnosed based on RIFLE creatinine criteria within 72 hours postoperatively. Serum creatinine is measured preoperatively, on the day of the surgery, and 1st, 2nd, and 3rd postoperative days.
5. Methods

   * Patients are randomized into 2 groups (Desflurane group and Sevoflurane group) depending on the agent administered during anesthesia
   * For the quantitative analysis for subclinical AKI, urine interleukin-6 (IL-6), plasma and urine neutrophil gelatinase-associated lipocalin (NGAL), serum cystatin C, urine liver-type fatty acid-binding protein (L-FABP), urine N-acetyl-β-D-Glucosaminidase (NAG), and urine albumin concentration are measured preoperatively, on the day of the surgery, and 1st postoperative day.
   * Demographic data, preoperative medication, past medical history, perioperative data related to anesthesia and surgery, and data related to outcome are also sampled.
   * Postoperative clinical course is followed until the patients are discharged.
   * Incidence rate of postoperative AKI and biomarkers are compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Forty adult patients (20 patients in each group) who are planned to undergo liver resection surgery are included.

Exclusion Criteria:

* Patients who undergo less invasive resection surgery under thoracoscopy or laparoscopy are excluded. Patients with chronic kidney disease, or allergic to any anesthetic agents used in the study are also excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | within 72 hours postoperatively
  Postoperative acute kidney injury is defined based on RIFLE creatinine criteria.

SECONDARY OUTCOMES:
Urine IL-6 concentration | On the day of surgery and postoperative day 1
  Urine IL-6 concentration is measured pre- and postoperatively to detect subclinical acute kidney injury.
Plasma NGAL concentration | On the day of surgery and postoperative day 1
  Plasma NGAL concentration is measured pre- and postoperatively to detect subclinical acute kidney injury.
Urine NGAL concentration | On the day of surgery and postoperative day 1
  Urine NGAL concentration is measured pre- and postoperatively to detect subclinical acute kidney injury.
Serum cystatin C concentration | On the day of surgery and postoperative day 1
  Serum cystatin C concentration is measured pre- and postoperatively to detect subclinical acute kidney injury.
Urine L-FABP concentration | On the day of surgery and postoperative day 1
  Urine L-FABP concentration is measured pre- and postoperatively to detect subclinical acute kidney injury.
Urine NAG concentration | On the day of surgery and postoperative day 1
  Urine NAG concentration is measured pre- and postoperatively to detect subclinical acute kidney injury.
Urine albumin concentration | On the day of surgery and postoperative day 1
  Urine albumin concentration is measured pre- and postoperatively to detect subclinical acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Koshi Makita, M.D., Principal Investigator — Tokyo Medical and Dental University
Locations (1):
- Tokyo Medical and Dental University, Tokyo, Japan